CLINICAL TRIAL: NCT06617052
Title: Efficacy and Safety of Preoperative (Chemo)Radiotherapy for Locally Recurrent Rectal Cancer: A Prospective, Single-arm Observational Study
Brief Title: Preoperative (Chemo)Radiotherapy for Locally Recurrent Rectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024ZSLYEC-487
Record Dates: First submitted 2024-09-18; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Locally Recurrent Rectal Cancer; Preoperative Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through an observational study, the efficacy and safety of preoperative chemoradiotherapy followed by surgery in patients with recurrent rectal cancer were assessed. The primary population included patients with (potentially) resectable locally recurrent rectal cancer, excluding those with distant metastases. The study design was a prospective, open-label, single-arm observational study. The primary endpoint was the pCR (pathological complete response) rate, while secondary endpoints included R0 resection rate, local recurrence-free survival, overall survival, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* ECOG performance status of 0-1
* Histologically, cytologically, or MRI/contrast-enhanced CT confirmed pelvic recurrence. At least one measurable pelvic lesion according to RECIST 1.1
* No distant metastases outside the pelvis
* (Potentially) resectable lesion
* No history of radiotherapy within the 6 months prior to enrollment
* No prior chemotherapy; or received postoperative adjuvant therapy but not systemic chemotherapy for metastatic lesions
* Investigator-assessed life expectancy of at least 24 weeks
* Adequate organ function (bone marrow, liver, kidney, and coagulation function) demonstrated within 7 days prior to the first dose, without the use of blood products or hematopoietic growth factors
* Not pregnant or breastfeeding. Effective contraception must be used during the study and for 6 months after the last dose
* Fully informed and willing to provide written informed consent to participate in the trial

Exclusion Criteria:

* Severe electrolyte abnormalities
* Active coronary artery disease, severe/unstable angina, newly diagnosed angina, or myocardial infarction within 12 months prior to study participation Thromboembolic events such as cerebrovascular accidents (including transient ischemic attacks), pulmonary embolism, or deep vein thrombosis within the past 6 months
* New York Heart Association (NYHA) class II or higher congestive heart failure
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); untreated active hepatitis (hepatitis B defined as HBV-DNA ≥ 500 IU/ml, or hepatitis C defined as HCV-RNA above the detection limit of the assay) or co-infection with hepatitis B and C
* Active inflammatory bowel disease or other colorectal diseases causing chronic diarrhea
* Any active, known, or suspected autoimmune disease. Stable conditions not required systemic immunosuppressive therapy are allowed, such as type I diabetes, hypothyroidism requiring only hormone replacement therapy, and skin conditions (e.g., vitiligo, psoriasis, and alopecia) not requiring systemic treatment
* Interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, or acute pneumonia)
* Known or suspected history of allergy to any study-related medications
* Clinically detectable second primary malignancy or history of another malignancy within the past 5 years
* Pregnant or breastfeeding women, or women with a positive pregnancy test before the first dose, or female participants and their partners unwilling to use strict contraception during the study
* Any clinical or laboratory abnormalities or compliance issues that the investigator deems unsuitable for study participation
* Severe psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: locally recurrent rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-19 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response | up to 26 weeks
  The resected tumor tissue and regional lymph nodes were pathologically assessed, revealing no residual tumor cells. The tumor lesions had completely disappeared, and no new lesions were detected.

SECONDARY OUTCOMES:
R0 rates | up to 26 weeks
  The complete tumor resection rate is defined as the absence of cancer cells at the resection margins under a microscope, with no visible or microscopic residual cancer cells, indicating that the lesion has been entirely removed.
progression-free survival | 5 years
  The interval between the start of enrollment and local recurrence, progression of local recurrence, distant metastasis, or death.
overall survival | 5 years
  The interval between the start of enrollment and death.

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China